CLINICAL TRIAL: NCT00700596
Title: Psychotomimetic Effects of Kappa Opioid Receptor Agonist Salvinorin A in Healthy Controls
Brief Title: Effects of Salvinorin A in Healthy Controls
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Principal Investigator, Mohini Ranganathan, Associate Professor of Psychiarty, Yale University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 0707002884
Record Dates: First submitted 2008-06-13; First posted 2008-06-18 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Healthy
Keywords: Salvia; SA; Salvinorin; Psychotomimetic Effects
MeSH Terms: interventions — salvinorin A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Active Comparator): Salvinorin A (SA)
  Interventions: Drug: Salvinorin A
- 2 (Placebo Comparator): Control or Placebo SA
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Salvinorin A — Low dose: Active SA 250μg Medium Dose: Active SA 500μg High Dose: Active SA 750μg
  Other Names: SA; Salvia; Salvia Divinorim
  Arms: 1
Drug: Placebo — Control or Placebo SA (30 % ethanolic solution)
  Arms: 2

SUMMARY:
This study evaluates the effects of Salvinorin A (SA). SA is the active ingredient of the plant Salvia divinorum that is known to have been used by Mexican Indians as part of religious rituals. The purpose of this project is to understand what people experience when they consume Salvinorin A.

ELIGIBILITY:
Inclusion Criteria:

-Previous exposure to inhaled Salvinorin A (SA).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2009-02-12 (Actual); Primary Completion 2014-08-22 (Actual); Study Completion 2014-08-22 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale, Clinician Administered Dissociative Symptoms Scale, Visual Analog Scale, Assessment of Opioid Effects, Cognitive Testing | Time Frame: -30, +10, +30, +90, +120. +200

CONTACTS AND LOCATIONS:
Overall Officials: Mohini Ranganathan, M.D., Principal Investigator — Yale University School of Medicine, Dept of Psychiatry
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States